CLINICAL TRIAL: NCT03443076
Title: A Randomized, Crossover Study to Assess the Relative Bioavailability of Eicosapentaenoic Acid and Docosahexaenoic Acid in a Self-micro-emulsifying Delivery System (SMEDS) Formulation Compared With a Standard Omega-3-acid Ethyl Ester Product
Brief Title: Bioavailability of EPA + DHA in a SMEDS Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Pharmavite LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MB-1705
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Bioavailability
MeSH Terms: interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPA + DHA in SMEDS Formulation (Experimental): Subject will receive a single 500 mg oral dose of EPA + DHA in a SMEDS formulation
  Interventions: Dietary Supplement: EPA + DHA in SMEDS Formulation
- EPA + DHA (Lovaza) (Active Comparator): Subject will receive a single 840 mg oral dose of EPA + DHA as Lovaza
  Interventions: Other: Lovaza (active comparator; already FDA approved)

INTERVENTIONS:
Dietary Supplement: EPA + DHA in SMEDS Formulation — A single dose of 500 mg EPA + DHA administered in a self-micro-emulsifying delivery system (SMEDS) formulation
  Arms: EPA + DHA in SMEDS Formulation
Other: Lovaza (active comparator; already FDA approved) — A single dose of 840 mg EPA + DHA administered as Lovaza. This intervention was used as an active comparator in this study. Lovaza was already FDA-approved when the study was conducted.
  Arms: EPA + DHA (Lovaza)

SUMMARY:
This study will assess the relative bioavailability of 500 mg eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) in a self-micro-emulsifying delivery system (SMEDS) formulation compared with a standard omega-3-acid ethyl ester product in healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.50-29.99 kg/m2
* Good health on basis of medical history and routine laboratory tests
* Score of at least 7 on vein access scale
* Willing and able to remain at site for extended testing periods, including a total of 4 overnight stays, and to consume foods and products provided by study staff on those days
* Willing to abstain from alcohol for 24 h prior to clinic admission
* No plans to change smoking habits or other nicotine use
* Willing to undergo 13 venipunctures during each treatment period

Exclusion Criteria:

* Screening lab test of clinical significance
* Positive urine drug screen
* Clinically significant endocrine, cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic, gastrointestinal or biliary disorder
* Uncontrolled hypertension
* Recent history or presence of cancer
* Difficulty swallowing capsules
* Recent blood donation or blood loss
* Recent consumption of high-dose fish oil or fish
* Recent use of any prescribed medication or over-the-counter medicinal products, including herbal or dietary supplements (except daily omega-3 fatty acid-free vitamin and/or mineral supplement or occasional use of acetaminophen or non-steroidal anti-inflammatory drugs)
* Signs or symptoms of active infection or has recently taken antibiotics
* Recent history or strong potential for drug or alcohol abuse
* Pregnant, planning to be pregnant during the study, lactating or of childbearing potential and unwilling to commit to use of a medically approved form of contraception throughout the study (note: hormonal contraceptive use is not allowed)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted, dose-normalized geometric mean ratio for SMEDS/Lovaza for EPA + DHA area under the curve (AUC) 0-24 hours | 0-24 h on Days 0-1 and on Days 14-15

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research, LLC
Locations (2):
- United States (2):
  - MB Clinical Research, LLC, Boca Raton, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maki KC, Palacios OM, Buggia MA, Trivedi R, Dicklin MR, Maki CE. Effects of a Self-micro-emulsifying Delivery System Formulation Versus a Standard omega-3 Acid Ethyl Ester Product on the Bioavailability of Eicosapentaenoic Acid and Docosahexaenoic Acid: A Study in Healthy Men and Women in a Fasted State. Clin Ther. 2018 Dec;40(12):2065-2076. doi: 10.1016/j.clinthera.2018.10.014. Epub 2018 Nov 16. PMID 30454850